CLINICAL TRIAL: NCT03442985
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Palovarotene in Subjects With Multiple Osteochondromas
Brief Title: An Efficacy and Safety Study of Palovarotene for the Treatment of MO
Acronym: MO-Ped
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial was terminated early to analyze the accumulated data and evaluate the efficacy, safety and future of palovarotene in MO.
Sponsor: Clementia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PVO-2A-201; 2017-002751-28 (EudraCT Number)
Record Dates: First submitted 2017-10-11; First posted 2018-02-22 (Actual); Results first posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Exostoses, Multiple Hereditary
Keywords: Multiple osteochondromas; Osteochondroma; Palovarotene; Hereditary multiple exostoses; HME; MO; Retinoic acid receptor gamma agonist; Retinoic acid receptor agonist
MeSH Terms: conditions — Exostoses, Multiple Hereditary; Osteochondroma | interventions — Palovarotene

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Palovarotene 2.5 mg daily regimen (Experimental)
  Interventions: Drug: Palovarotene 2.5 mg
- Palovarotene 5.0 mg daily regimen (Experimental)
  Interventions: Drug: Palovarotene 5.0 mg
- Placebo regimen (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Palovarotene 2.5 mg — Subjects received a weight-adjusted dose equivalent of 2.5 mg palovarotene, once daily, for up to 24 months.
  Arms: Palovarotene 2.5 mg daily regimen
Drug: Palovarotene 5.0 mg — Subjects received a weight-adjusted dose equivalent of 5.0 mg palovarotene, once daily, for up to 24 months.
  Arms: Palovarotene 5.0 mg daily regimen
Other: Placebo — Subjects received placebo, once daily, for up to 24 months.
  Arms: Placebo regimen

SUMMARY:
This is a randomized, double-blind, placebo-controlled study comparing the safety and efficacy of 2 dosage regimens of palovarotene versus placebo in preventing disease progression in pediatric subjects with multiple osteochondromas (MO).

DETAILED DESCRIPTION:
Multiple osteochondromas is a rare condition where children develop multiple benign cartilage-capped bony tumors called osteochondromas on bones throughout the body, resulting in pain, deformity, limb length discrepancy, disability, and eventually arthritis and possible malignancy. The primary objective is to compare the efficacy of two dosage regimens of palovarotene with placebo to prevent the formation of new osteochondromas in pediatric MO subjects with exostosin 1 or exostosin 2 gene mutations. Osteochondroma formation was assessed by whole body magnetic resonance imaging (MRI). Secondary efficacy objectives were to compare the effects of palovarotene with placebo on the volume of osteochondromas as assessed by MRI; the proportion of subjects with no new osteochondromas as assessed by whole-body MRI; the annualized rate of new or worsening deformities; the annualized rate of MO-related surgeries; and palatability. The overall safety and pharmacokinetics of palovarotene and the effects of palovarotene on linear growth, bone growth plates, bone mineral density, quality of life, and pain due to osteochondromas was also studied.

ELIGIBILITY:
Key Inclusion Criteria:

* Written, signed, and dated informed subject/parent consent and age-appropriate assent (performed according to local regulations).
* A clinical diagnosis of MO with disease-causing exostosin 1 or 2 gene mutations.
* Male or female from 2 to 14 years of age.
* Female subjects must be premenarchal at screening.
* A bone age at screening of 14 years or less.
* Symptomatic MO, defined as five or more clinically evident osteochondromas and a new or enlarged osteochondroma that occurred in the preceding 12 months, five or more clinically evident osteochondromas and the presence of a painful osteochondroma, a skeletal deformity, a joint limitation, or prior surgery for a MO-related complication.
* The ability to undergo whole body MRI with or without sedation/general anesthesia.
* Use of two effective methods of birth control during treatment, and for 1 month after treatment discontinuation, unless committed to true abstinence from heterosexual sex. Sexually active females of child-bearing potential must also agree to start effective methods of birth control at screening.

Key Exclusion Criteria:

* Weight under 10 kg.
* Other syndromic conditions such as Langer-Giedion or Potocki-Shaffer.
* Any subject with neurologic signs suggestive of spinal cord impingement.
* Concomitant medications that are strong inhibitors or inducers of cytochrome P450 3A4 activity.
* Amylase or lipase >2 times the above the upper limit of normal (>2×ULN) or with a history of chronic pancreatitis.
* Elevated aspartate aminotransferase or alanine aminotransferase above 2.5×ULN.
* Any surgical implant that is contraindicated for MRI.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (31):
- United States (13):
  - Children's Orthopaedic Center, Los Angeles, California
  - Shriners Hospital for Children - Sacramento, Sacramento, California
  - University of California-San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - The Paley Institute, West Palm Beach, Florida
  - Shriners Hospital for Children - Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Shriners Hospitals for Children - Portland, Portland, Oregon
  - The Children's Hospital of Philadelphia (CHOP), Philadelphia, Pennsylvania
  - Shriners Hospital for Children - Philadelphia, Philadelphia, Pennsylvania
  - Memorial Hermann Hospital, Houston, Texas
- Westmead Children's Hospital, Westmead, New South Wales, Australia
- UZ Antwerpen, Edegem, Antwerp, Belgium
- Canada (3):
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Shriners Hospital for Children - Canada, Montreal, Quebec
- France (2):
  - Hôpital universitaire Necker - Enfants Malades, Paris
  - Hôpital des Enfants, CHU de Toulouse, Toulouse
- Istituti Ortopedici Rizzoli, Bologna, Emilia-Romagna, Italy
- Japan (2):
  - Nagoya University Hospital, Nagoya, Aiti
  - Osaka University Hospital, Suita, Osaka
- OLVG locatie Oost, Amsterdam, North Holland, Netherlands
- Hospital Pediátrico de Coimbra, Coimbra, Portugal
- Hospital Universitario La Paz, Madrid, Spain
- Turkey (Türkiye) (2):
  - Ege University Medical Faculty Hospital, Bornova, İzmir
  - Bezmialem Vakif University Medical Faculty Hospital, Istanbul
- United Kingdom (3):
  - Evelina London Children's Hospital, London
  - Royal Manchester Childrens Hospital, Manchester
  - Royal National Orthopaedic Hospital, Stanmore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inubushi T, Lemire I, Irie F, Yamaguchi Y. Palovarotene Inhibits Osteochondroma Formation in a Mouse Model of Multiple Hereditary Exostoses. J Bone Miner Res. 2018 Apr;33(4):658-666. doi: 10.1002/jbmr.3341. Epub 2017 Nov 30. PMID 29120519
- [Derived] Sangiorgi L, Conrad EU, Shih F, Strahs A, Feldman DS. Palovarotene for patients with multiple hereditary exostosis: results of MO-Ped, a terminated, randomized, placebo-controlled, double-blind phase 2 trial. Sci Rep. 2025 Nov 4;15(1):38563. doi: 10.1038/s41598-025-22554-6. PMID 41188357
- See also: MHE Coalition — http://www.mhecoalition.org/
- See also: MHE Research Foundation — http://www.mherf.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 2 placebo-controlled study was conducted in pediatric participants with multiple osteochondromas (MO) at 29 study sites in 11 countries between 22 March 2018 and 30 October 2020. For sites in the European Union, participants from 7 to <15 years of age were enrolled first and participants from 2 to <7 years of age were enrolled after the 6-month bone safety data from at least 20 skeletally immature participants.
Pre-assignment Details: Study consisted of a screening period (up to 35 days), followed by a double-blind treatment period (24 months) and safety follow-up period (6 months). Participants were randomized in a 1:1:1 ratio to palovarotene 2.5 milligram (mg) or 5.0 mg or placebo. A total of 193 participants received at least 1 dose of study drug and were included in the study analysis.
Groups:
- Placebo: Participants were to receive placebo matching with palovarotene capsules orally once daily, for up to 24 months.
- Palovarotene 2.5 mg: Participants were to receive weight-adjusted dose equivalent of palovarotene 2.5 mg capsules orally once daily, for up to 24 months.
- Palovarotene 5.0 mg: Participants were to receive weight-adjusted dose equivalent of palovarotene 5.0 mg capsules orally once daily, for up to 24 months.
Period: Overall Study
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Started (Received treatment) | 62 | 66 | 65
Completed | 0 | 0 | 0
Not Completed | 62 | 66 | 65
Not completed — Sponsor Request | 55 | 60 | 54
Not completed — Lost to Follow-up | 5 | 2 | 7
Not completed — Withdrawal by Subject | 2 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Safety set included randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg | Total
Number analyzed (Participants) | 62 | 66 | 65 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.9 (2.5) | 7.8 (3.1) | 7.4 (3.1) | 7.7 (2.9)
Age, Customized [Count of Participants; unit: Participants]
  2 to 5 years | 13 | 17 | 19 | 49
  6 to 10 years | 38 | 33 | 35 | 106
  11 to 14 years | 11 | 16 | 11 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 27 | 76
  Male | 39 | 40 | 38 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 50 | 52 | 150
  Black Or African American | 0 | 2 | 2 | 4
  Asian | 5 | 3 | 3 | 11
  American Indian Or Alaska Native | 0 | 1 | 0 | 1
  Multiple | 6 | 7 | 5 | 18
  Other | 0 | 0 | 1 | 1
  Missing | 3 | 3 | 2 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 7 | 20
  Not Hispanic or Latino | 56 | 58 | 57 | 171
  Missing | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of New Osteochondromas (OCs)
Description: The annualized rate of new OCs was assessed by whole-body magnetic resonance imaging (MRI) (that is, the total number of new OCs divided by the time in years between the baseline and latest post-baseline MRI).
Time Frame: Month 12
Population: The Full Analysis Set (FAS) included randomized participants who received at least 1 dose of study drug. Only data from the 56 participants for whom Month 12 efficacy imaging data were available were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of new OCs per year
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 16 | 17 | 23
number of new OCs per year | 0.119 [0.031 to 0.461] | 0.363 [0.148 to 0.888] | 0.172 [0.073 to 0.404]
Statistical Analysis 1: Comparison: Palovarotene 2.5 mg vs Palovarotene 5.0 mg; Palovarotene 2.5 mg versus (vs) Palovarotene 5.0 mg: The annualized rate for number of new OCs was estimated using an unadjusted negative binomial regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.2556, Negative binomial regression model — The p-values were not adjusted for multiple testing due to small sample size; Risk Ratio (RR) = 2.109, 95% CI 2-sided [0.583 to 7.638]
Statistical Analysis 2: Comparison: Placebo vs Palovarotene 2.5 mg; Palovarotene 2.5 mg vs Placebo: The annualized rate for number of new OCs was estimated using an unadjusted negative binomial regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.1788, Negative binomial regression model — The p-values were not adjusted for multiple testing due to small sample size; Risk Ratio (RR) = 3.040, 95% CI 2-sided [0.601 to 15.373]
Statistical Analysis 3: Comparison: Placebo vs Palovarotene 5.0 mg; Palovarotene 5.0 mg vs Placebo: The annualized rate for number of new OCs was estimated using an unadjusted negative binomial regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.6570, Negative binomial regression model — The p-values were not adjusted for multiple testing due to small sample size; Risk Ratio (RR) = 1.441, 95% CI 2-sided [0.287 to 7.234]

2. Secondary Outcome: Mean Change From Baseline in the Total Volume of New OCs at Month 12
Description: The change from baseline in the total volume of OCs was assessed by whole-body MRI. Baseline was defined as the last available value prior to first administration of study drug.
Time Frame: Baseline (Day 1) and Month 12
Population: The FAS included randomized participants who received at least 1 dose of study drug. Only data from the 56 participants for whom Month 12 efficacy imaging data were available were included in the analysis.
Measure: Mean (Standard Deviation); unit: cubic millimeter
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 16 | 17 | 23
cubic millimeter | 10476.7 (23294.9) | 5250.5 (11754.7) | 10911.0 (35869.6)
Statistical Analysis 1: Comparison: Palovarotene 2.5 mg vs Palovarotene 5.0 mg; Palovarotene 2.5 mg vs Palovarotene 5.0 mg: The mean difference in the change from baseline for total OC volume was estimated using an unadjusted estimation equation model with independent working covariance matrix to address potential correlation within the same family members; Test type: Other; p = 0.4252, Unadjusted estimation equation model — The p-values were not adjusted for multiple testing due to small sample size; Risk Ratio (RR) = -4412.6, 95% CI 2-sided [-15257.3 to 6432.1]
Statistical Analysis 2: Comparison: Placebo vs Palovarotene 2.5 mg; Palovarotene 2.5 mg vs Placebo: The mean difference in the change from baseline for total OC volume was estimated using an unadjusted estimation equation model with independent working covariance matrix to address potential correlation within the same family members; Test type: Other; p = 0.4053, Unadjusted estimation equation model — The p-values were not adjusted for multiple testing due to small sample size; Risk Ratio (RR) = -4640.9, 95% CI 2-sided [-15570.8 to 6289.0]
Statistical Analysis 3: Comparison: Placebo vs Palovarotene 5.0 mg; Palovarotene 5.0 mg vs Placebo: The mean difference in the change from baseline for total OC volume was estimated using an unadjusted estimation equation model with independent working covariance matrix to address potential correlation within the same family members; Test type: Other; p = 0.9677, Unadjusted estimation equation model — The p-values were not adjusted for multiple testings due to small sample size; Risk Ratio (RR) = -228.3, 95% CI 2-sided [-11265.0 to 10808.4]

3. Secondary Outcome: Percentage of Participants With No New OCs
Description: The percentage of participants with no new OCs as assessed by whole-body MRI. Participants with new OCs not identified by MRI due to surgical resection during the treatment period were categorized as having new OCs for this analysis.
Time Frame: Month 12
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 16 | 17 | 23
percentage of participants | 62.5 | 47.1 | 56.5
Statistical Analysis 1: Comparison: Palovarotene 2.5 mg vs Palovarotene 5.0 mg; Test type: Other; p = 0.5025, Regression, Logistic; Logistic regression was adjusted for the following covariates: baseline age, sex, and Ext1/2 mutation status; Odds Ratio (OR) = 0.643, 95% CI 2-sided [0.177 to 2.335]
Statistical Analysis 2: Comparison: Placebo vs Palovarotene 2.5 mg; Test type: Other; p = 0.3763, Regression, Logistic; Logistic regression was adjusted for the following covariates: baseline age, sex, and Ext1/2 mutation status; Odds Ratio (OR) = 0.528, 95% CI 2-sided [0.128 to 2.175]
Statistical Analysis 3: Comparison: Placebo vs Palovarotene 5.0 mg; Test type: Other; p = 0.7714, Regression, Logistic; Logistic regression was adjusted for the following covariates: baseline age, sex, and Ext1/2 mutation status; Odds Ratio (OR) = 0.820, 95% CI 2-sided [0.215 to 3.123]

4. Secondary Outcome: Annualized Rate of New or Worsening Deformities
Description: The annualized rate of new or worsening deformities as assessed by radiographic imaging of both upper and lower limbs.
Time Frame: Month 12
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: number of deformities per year
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 16 | 18 | 22
number of deformities per year | 1.797 [1.272 to 2.537] | 1.802 [1.209 to 2.684] | 1.895 [1.584 to 2.266]
Statistical Analysis 1: Comparison: Palovarotene 2.5 mg vs Palovarotene 5.0 mg; Palovarotene 2.5 mg vs Palovarotene 5.0 mg: The annualized rate for number of new or worsening deformities was estimated using an unadjusted negative binomial regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.8155, Negative binomial regression model — The p-values were not adjusted for multiple testing due to small sample size. The correlation matrix type = compound symmetry was used; Risk Ratio (RR) = 0.951, 95% CI 2-sided [0.623 to 1.451]
Statistical Analysis 2: Comparison: Placebo vs Palovarotene 2.5 mg; Palovarotene 2.5 mg vs Placebo: The annualized rate for number of new or worsening deformities was estimated using an unadjusted negative binomial regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.9918, Negative binomial regression model — [p-value comment as in outcome 4, analysis 1]; Risk Ratio (RR) = 1.003, 95% CI 2-sided [0.592 to 1.699]
Statistical Analysis 3: Comparison: Placebo vs Palovarotene 5.0 mg; Palovarotene 5.0 mg vs Placebo: The annualized rate for number of new or worsening deformities was estimated using an unadjusted negative binomial regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.7997, Negative binomial regression model — [p-value comment as in outcome 4, analysis 1]; Risk Ratio (RR) = 1.055, 95% CI 2-sided [0.700 to 1.589]

5. Secondary Outcome: Annualized Rate of MO-Related Surgeries
Description: The MO-related surgeries included any procedure indicated for the treatment of MO, such as an excision of a symptomatic OC or correction of a limb deformity.
Time Frame: Month 12
Population: The FAS included randomized participants who received at least 1 dose of study drug. Participants with planned surgeries within 6 months of enrollment to remove symptomatic OCs or to correct deformities present at baseline, and/or had surgical procedures that were a continuation of a previous procedure were excluded in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: number of MO-related surgeries per year
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 4 | 8 | 7
number of MO-related surgeries per year | 2.087 [1.099 to 3.964] | 3.454 [1.850 to 6.451] | 2.231 [1.638 to 3.038]
Statistical Analysis 1: Comparison: Palovarotene 2.5 mg vs Palovarotene 5.0 mg; Palovarotene 2.5 mg vs Palovarotene 5.0 mg: The annualized rate for number of MO-related surgeries was estimated using an unadjusted poisson regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.2186, Poisson regression model — The p-values were not adjusted for multiple testing due to small sample size. The correlation matrix type = independent was used; Risk Ratio (RR) = 1.548, 95% CI 2-sided [0.772 to 3.108]
Statistical Analysis 2: Comparison: Placebo vs Palovarotene 2.5 mg; Palovarotene 2.5 mg vs Placebo: The annualized rate for number of MO-related surgeries was estimated using an unadjusted poisson regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.2700, Poisson regression model — [p-value comment as in outcome 5, analysis 1]; Risk Ratio (RR) = 1.655, 95% CI 2-sided [0.676 to 4.052]
Statistical Analysis 3: Comparison: Placebo vs Palovarotene 5.0 mg; Palovarotene 5.0 mg vs Placebo: The annualized rate for number of MO-related surgeries was estimated using an unadjusted poisson regression model, offsetted by log-transformed follow-up time (years) to obtain annualized rate; Test type: Other; p = 0.8546, Poisson regression model — [p-value comment as in outcome 5, analysis 1]; Risk Ratio (RR) = 1.069, 95% CI 2-sided [0.524 to 2.178]

6. Secondary Outcome: Maximum Observed Plasma Drug Concentrations at Steady State (Cmax,ss) of Palovarotene
Description: The Cmax,ss of palovarotene was evaluated. The pharmacokinetic (PK) sampling was performed at Month 1. If samples could not be obtained at Month 1, then one additional attempt was made at a subsequent visit.
Time Frame: Month 1: pre-dose and 3, 6, 10 and 24 hours post-dose
Population: The Pharmacokinetic Set (PKS) included participants receiving treatment with palovarotene and with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 49 | 52
nanogram per milliliter (ng/mL) | 18.0 (50.2) | 34.9 (63.3)

7. Secondary Outcome: Minimum Observed Plasma Drug Concentrations at Steady State (Cmin,ss) of Palovarotene
Description: The Cmin,ss of palovarotene was evaluated. The PK sampling was performed at Month 1. If samples could not be obtained at Month 1, then one additional attempt was made at a subsequent visit.
Time Frame: Month 1: pre-dose and 3, 6, 10 and 24 hours post-dose
Population: The PKS included participants receiving treatment with palovarotene and with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 49 | 53
ng/mL | 0.314 (86.1) | 0.674 (83.3)

8. Secondary Outcome: Time to Maximum Observed Drug Concentration at Steady State (Tmax,ss) of Palovarotene
Description: The Tmax,ss of palovarotene was evaluated. The PK sampling was performed at Month 1. If samples could not be obtained at Month 1, then one additional attempt was made at a subsequent visit.
Time Frame: Month 1: pre-dose and 3, 6, 10 and 24 hours post-dose
Population: The PKS included participants receiving treatment with palovarotene and with evaluable PK data.
Measure: Median (Full Range); unit: hour
Arm/Group | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 49 | 52
hour | 3.00 [2.47 to 10.00] | 3.01 [2.42 to 24.25]

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve at Steady State From Time 0 to 24 Hours After Dosing (AUC0-24,ss) of Palovarotene
Description: The AUC0-24,ss of palovarotene was evaluated. The PK sampling was performed at Month 1. If samples could not be obtained at Month 1, then one additional attempt was made at a subsequent visit.
Time Frame: Month 1: pre-dose and 3, 6, 10 and 24 hours post-dose
Population: The PKS included participants receiving treatment with palovarotene and with evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 47 | 46
hour*ng/mL | 112 (29.1) | 241 (42.7)

10. Secondary Outcome: Number of Participants With Palatability of Sprinkled Palovarotene and Placebo
Description: Palatability of palovarotene and placebo when sprinkled on specific foods as assessed with a 5-point hedonic face scale at the first dose (Day 1) and at Month 1 in all participants (including <4 years old) who sprinkled the palovarotene or placebo onto a spoonful of specific foods. The hedonic face scale ranges from 1 to 5 where, 1= dislike very much, 2= dislike slightly, 3= neither like nor dislike, 4= like slightly, 5= like very much. Higher scores indicate positive outcome.
Time Frame: Day 1 and Month 1
Population: The Safety set included randomized participants who received at least 1 dose of study drug. Only data from the participants analyzed at Day 1 and Month 1 were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
Number analyzed (Participants) | 21 | 15 | 11
Participants
  Day 1: Dislike very much | 0 | 1 | 0
  Day 1: Dislike a little | 1 | 1 | 0
  Day 1: Not sure | 6 | 3 | 3
  Day 1: Like a little | 3 | 5 | 3
  Day 1: Like very much | 11 | 5 | 5
  Month 1: Dislike very much | 1 | 0 | 0
  Month 1: Dislike a little | 1 | 1 | 1
  Month 1: Not sure | 5 | 1 | 3
  Month 1: Like a little | 8 | 5 | 1
  Month 1: Like very much | 6 | 8 | 6

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were to be collected from the start of the first study drug (Day 1) up to 7 days after last study drug intake, assessed until data cut-off for study termination (maximum of 595 days).
Description: The Safety set included randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Palovarotene 2.5 mg | Palovarotene 5.0 mg
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/66 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/62 | 2/66 | 2/65
Other Adverse Events (participants affected / at risk) | 41/62 | 56/66 | 56/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=62) | Palovarotene 2.5 mg (N=66) | Palovarotene 5.0 mg (N=65)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Status Epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=62) | Palovarotene 2.5 mg (N=66) | Palovarotene 5.0 mg (N=65)
Rash (Skin and subcutaneous tissue disorders) | 7 (12) | 17 (31) | 25 (50)
Dry Skin (Skin and subcutaneous tissue disorders) | 7 (9) | 16 (19) | 19 (23)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7) | 8 (9) | 7 (9)
Rash Generalised (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3) | 5 (5)
Lip Dry (Gastrointestinal disorders) | 3 (3) | 6 (6) | 11 (11)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (4) | 7 (9)
Dry Mouth (Gastrointestinal disorders) | 3 (3) | 4 (4) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 9 (9)
Headache (Nervous system disorders) | 6 (8) | 4 (4) | 3 (4)

LIMITATIONS AND CAVEATS:
The Sponsor terminated the study early due to a partial clinical hold instituted by the Food and Drug Administration. Recruitment was stopped before full enrollment was reached, and study drug administration was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03442985/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03442985/SAP_001.pdf